CLINICAL TRIAL: NCT01388491
Title: A Multinational, Multicenter, Randomized, Open-Label Study to Evaluate the Impact of DR-102 Compared to a 28-day Standard Oral Contraceptive Regimen, on Hemosatic Parameters in Healthy Women
Brief Title: A Multinational Study to Evaluate the Effects of a 28-Day Oral Contraceptive on Hemostatic Parameters in Healthy Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DSG-HSP-201
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Results first posted 2013-11-27 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Hemostasis; Oral Contraceptive
Keywords: Contraception; Hemostasis; Blood Coagulation
MeSH Terms: conditions — Thrombosis | interventions — Desogestrel; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment I: (DR-102) (Experimental): 21 days of combination active pills (containing 150 mcg desogestrel [DSG]/20 mcg ethinyl estradiol [EE]), followed by 7 days of 10 mcg EE, taken orally for 6 consecutive 28-day cycles
  Interventions: Drug: desogestrel/ethinyl estradiol and ethinyl estradiol
- Treatment II (Active Comparator): 21 days combination active pills (containing 150 mcg DSG/20 mcg EE), taken orally and followed by 7 days of no treatment for a total of 6 consecutive 28-day cycles
  Interventions: Drug: desogestrel/ethinyl estradiol

INTERVENTIONS:
Drug: desogestrel/ethinyl estradiol and ethinyl estradiol
  Arms: Treatment I: (DR-102)
Drug: desogestrel/ethinyl estradiol
  Arms: Treatment II

SUMMARY:
This study is being conducted to evaluate the impact of DR-102, a 28-day oral contraceptive compared to a standard 28-day oral contraceptive regimen on hemostatic parameters in healthy women.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal, non-pregnant, non-lactating women age 18-40 years old
* Body Mass Index (BMI) ≥18 kg/m² and <30 kg/m²
* Regular spontaneous menstrual cycle
* Others as dictated by FDA-approved protocol

Exclusion Criteria:

* Any condition which contraindicates the use of combination oral contraceptives
* Any history of, or active, deep vein thrombosis, pulmonary embolism, or arterial thromboembolic disease within one year of screening
* Thrombophlebitis or thromboembolic disorders; known or suspected clotting disorders; thrombogenetic valvulopathies or rhythm disorders
* Others as dictated by FDA-approved protocol

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 293 (Actual)
Dates: Start 2011-10-31 (Actual); Primary Completion 2012-09-30 (Actual); Study Completion 2012-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Women's Health Research Protocol Chair, Study Chair — Teva Women's Health Research
Locations (27):
- Germany (6):
  - Teva Investigational Site 32064, Essen
  - Teva Investigational Site 32065, Frankfurt
  - Teva Investigational Site 32066, Frankfurt am Main
  - Teva Investigational Site 32062, Hamburg
  - Teva Investigational Site 32063, Hamburg
  - Teva Investigational Site 32061, Magdeburg
- Israel (6):
  - Teva Investigational Site 80013, Giv‘atayim
  - Teva Investigational Site 80015, Haifa
  - Teva Investigational Site 80017, Modiin
  - Teva Investigational Site 80014, RishonLe'zio
  - Teva Investigational Site 80018, Tel Aviv
  - Teva Investigational Site 80016, Tel Aviv
- Italy (7):
  - Teva Investigational Site 30014, Brescia
  - Teva Investigational Site 30009, Cagliari
  - Teva Investigational Site 30012, Catania
  - Teva Investigational Site 30013, Napoli
  - Teva Investigational Site 30010, Pavia
  - Teva Investigational Site 30007, Pisa
  - Teva Investigational Site 30016, Siena
- Spain (8):
  - Teva Investigational Site 31017, Barcelona
  - Teva Investigational Site 31015, Barcelona
  - Teva Investigational Site 31014, Barcelona
  - Teva Investigational Site 31016, Gava, Barcelona
  - Teva Investigational Site 31012, Lugo
  - Teva Investigational Site 31010, Madrid
  - Teva Investigational Site 31011, Madrid
  - Teva Investigational Site 31009, Vitoria-Gasteiz

REFERENCES:
- [Result] Peters K, Gordon N, Ricciotti N, Hsieh J, Howard B, Weiss H. Hemostatic effects of two desogestrel-containing combined oral contraceptive regimens: a multinational, multicenter, randomized, open-label study. Clin Exp Obstet Gynecol. 2016;43(3):334-40. PMID 27328486

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 351 healthy women screened for enrollment, 293 at 26 centers in the European Union (EU) (21 centers) and Israel (5 centers) met entry criteria and were considered to be eligible for this study.
Pre-assignment Details: Of the 58 women who were screened but not randomly assigned to receive treatment, 10 were excluded on the basis of inclusion/exclusion criteria, 32 withdrew consent, and 6 were lost to follow-up before the baseline visit. An additional 10 participants were not randomly assigned to treatment for other reasons.
Period: Overall Study
Arm/Group | Treatment I: (DR-102) | Treatment II
Started | 150 (number randomized) | 143
Safety Population | 145 (Safety: all randomized participants who took 1 or more doses of study drug) | 142
Intent-to-Treat (ITT) Population | 140 (ITT:participants in safety population with baseline (BL) + ≥1 post-BL prothrombin fragment 1+2 value) | 136
Per Protocol (PP) Population | 125 (PP: all data from ITT participants obtained prior to any major protocol violations) | 121
Completed | 116 | 114
Not Completed | 34 | 29
Not completed — Adverse Event | 10 | 9
Not completed — Sponsor Request | 9 | 7
Not completed — Withdrawal by Subject | 6 | 10
Not completed — Lost to Follow-up | 4 | 3
Not completed — Protocol Violation | 2 | 0
Not completed — Noncompliance | 2 | 0
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population (all randomized participants who took 1 or more doses of study drug)
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment I: (DR-102) | Treatment II | Total
Number analyzed (Participants) | 145 | 142 | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (4.98) | 27.0 (5.26) | 26.7 (5.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 142 | 287
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 140 | 136 | 276
  Black | 1 | 1 | 2
  Asian | 0 | 1 | 1
  American Indian or Alaskan Native | 0 | 1 | 1
  Other | 4 | 3 | 7
Weight [Mean (Standard Deviation); unit: kg] | 61.6 (10.35) | 60.1 (9.36) | 60.9 (9.89)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.9 (3.62) | 22.4 (3.06) | 22.6 (3.36)

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Change From Baseline Over the 6-Month Treatment Period in Prothrombin Fragment 1 + 2 Levels
Description: Normal range for this hemostatic parameter was 41 to 372 pmol/L. Participants were in a fasting state and had refrained from moderate to vigorous exercise prior to phlebotomy on the day of this lab draw. Change from baseline was analyzed using a repeated measures analysis of covariance with covariate adjustment for baseline, treatment, month, and the treatment by month interaction.
Time Frame: Baseline through Month 6
Population: Per-protocol (PP) population. PP population included all data from intent-to-treat (ITT) participants obtained prior to any major protocol violations. PP participants were analyzed according to the treatment actually received.
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Treatment I: (DR-102) | Treatment II
Number analyzed (Participants) | 125 | 121
pmol/L | 45.0 (15.24) | 56.8 (15.60)
Statistical Analysis 1: Comparison: Treatment I: (DR-102) vs Treatment II; Test type: Superiority or Other; p = 0.5892, ANCOVA — The p-value, least squares mean difference, and 95% CI for the treatment group comparison are based on a repeated measures ANCOVA with baseline, treatment, visit, and treatment-by-visit interaction as fixed factors, and subject as a random effect; Least Squares mean difference: Treatment I - Treatment II; Least Squares Mean Difference = -11.8, 95% CI 2-sided [-54.75 to 31.17]

2. Secondary Outcome: Least Squares Mean Change From Baseline Over the 6-Month Treatment Period in D-Dimer
Description: Normal range for this hemostatic parameter was 0 to 729 mcg/L. Participants were in a fasting state and had refrained from moderate to vigorous exercise prior to phlebotomy on the day of this lab draw. Change from baseline was analyzed using a repeated measures analysis of covariance with covariate adjustment for baseline, treatment, month, and the treatment by month interaction.
Time Frame: Baseline through Month 6
Population: Per protocol (PP) population with BL and at least 1 post-BL value for this measurement. PP population included all data from intent-to-treat (ITT) participants obtained prior to any major protocol violations. PP participants were analyzed according to the treatment actually received.
Measure: Least Squares Mean (Standard Error); unit: mcg/L
Arm/Group | Treatment I: (DR-102) | Treatment II
Number analyzed (Participants) | 118 | 114
mcg/L | 16.4 (10.29) | 13.4 (10.46)
Statistical Analysis 1: Comparison: Treatment I: (DR-102) vs Treatment II; Test type: Superiority or Other; p = 0.839, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares mean difference: Treatment I - Treatment II; Least Squares Mean Difference = 3.0, 95% CI 2-sided [-25.96 to 31.94]

3. Secondary Outcome: Least Squares Mean Change From Baseline Over the 6-Month Period in Protein S Total Antigen
Description: The normal range for this hemostatic parameter was 50% to 147%. Participants were in a fasting state and had refrained from moderate to vigorous exercise prior to phlebotomy on the day of this lab draw. Change from baseline was analyzed using a repeated measures analysis of covariance with covariate adjustment for baseline, treatment, month, and the treatment by month interaction.
Time Frame: Baseline through Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of normal 50% to 147%
Arm/Group | Treatment I: (DR-102) | Treatment II
Number analyzed (Participants) | 124 | 121
percentage of normal 50% to 147% | -11.4 (1.09) | -6.6 (1.10)
Statistical Analysis 1: Comparison: Treatment I: (DR-102) vs Treatment II; Test type: Superiority or Other; p = 0.0021, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares mean difference: Treatment I - Treatment II; Least Squares Mean Difference = -4.8, 95% CI 2-sided [-7.87 to -1.77]

4. Secondary Outcome: Least Squares Mean Change From Baseline Over the 6-Month Treatment Period in Protein C Activity
Description: The normal range for this hemostatic parameter was 70% to 180%. Participants were in a fasting state and had refrained from moderate to vigorous exercise prior to phlebotomy on the day of this lab draw. Change from baseline was analyzed using a repeated measures analysis of covariance with covariate adjustment for baseline, treatment, month, and the treatment by month interaction.
Time Frame: Baseline through Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of normal
Arm/Group | Treatment I: (DR-102) | Treatment II
Number analyzed (Participants) | 124 | 121
percentage of normal | 16.3 (1.90) | 13.0 (1.93)
Statistical Analysis 1: Comparison: Treatment I: (DR-102) vs Treatment II; Test type: Superiority or Other; p = 0.2312, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares mean difference: Treatment I - Treatment II; Least Squares Mean Difference = 3.2, 95% CI 2-sided [-2.08 to 8.58]

5. Secondary Outcome: Least Squares Mean Change From Baseline Over the 6-Month Treatment Period in Antithrombin
Description: Normal range for this hemostatic parameter was 75% to 130%. Participants were in a fasting state and had refrained from moderate to vigorous exercise prior to phlebotomy on the day of this lab draw. Change from baseline was analyzed using a repeated measures analysis of covariance with covariate adjustment for baseline, treatment, month, and the treatment by month interaction.
Time Frame: Baseline through Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of normal
Arm/Group | Treatment I: (DR-102) | Treatment II
Number analyzed (Participants) | 124 | 121
percentage of normal | -1.6 (1.17) | -3.2 (1.18)
Statistical Analysis 1: Comparison: Treatment I: (DR-102) vs Treatment II; Test type: Superiority or Other; p = 0.3440, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares mean difference: Treatment I - Treatment II; Least Squares Mean Difference = 1.6, 95% CI 2-sided [-1.70 to 4.85]

6. Secondary Outcome: Least Squares Mean Change From Baseline Over the 6-Month Treatment Period in Factor II Activity
Description: Normal range for this hemostatic parameter was 70% to 150%. Participants were in a fasting state and had refrained from moderate to vigorous exercise prior to phlebotomy on the day of this lab draw. Change from baseline was analyzed using a repeated measures analysis of covariance with covariate adjustment for baseline, treatment, month, and the treatment by month interaction.
Time Frame: Baseline through Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of normal
Arm/Group | Treatment I: (DR-102) | Treatment II
Number analyzed (Participants) | 118 | 114
percentage of normal | 3.3 (0.21) | 3.0 (0.21)
Statistical Analysis 1: Comparison: Treatment I: (DR-102) vs Treatment II; Test type: Superiority or Other; p = 0.2522, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares mean difference: Treatment I - Treatment II; Least Squares Mean Difference = 0.3, 95% CI 2-sided [-0.24 to 0.92]

7. Secondary Outcome: Least Squares Mean Change From Baseline Over the 6-Month Treatment Period in Factor VII
Description: Normal range for this hemostatic parameter was 60% to 150%. Participants were in a fasting state and had refrained from moderate to vigorous exercise prior to phlebotomy on the day of this lab draw. Change from baseline was analyzed using a repeated measures analysis of covariance with covariate adjustment for baseline, treatment, month, and the treatment by month interaction.
Time Frame: Baseline through Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of normal
Arm/Group | Treatment I: (DR-102) | Treatment II
Number analyzed (Participants) | 118 | 114
percentage of normal | 17.9 (0.81) | 15.1 (0.82)
Statistical Analysis 1: Comparison: Treatment I: (DR-102) vs Treatment II; Test type: Superiority or Other; p = 0.0143, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares mean difference: Treatment I - Treatment II; Least Squares Mean Difference = 2.9, 95% CI 2-sided [0.58 to 5.13]

8. Secondary Outcome: Least Squares Mean Change From Baseline Over the 6-Month Treatment Period in Factor VIII
Description: Normal range for this hemostatic parameter was 50% to 180%. Participants were in a fasting state and had refrained from moderate to vigorous exercise prior to phlebotomy on the day of this lab draw. Change from baseline was analyzed using a repeated measures analysis of covariance with covariate adjustment for baseline, treatment, month, and the treatment by month interaction.
Time Frame: Baseline through Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of normal
Arm/Group | Treatment I: (DR-102) | Treatment II
Number analyzed (Participants) | 118 | 114
percentage of normal | 11.1 (1.92) | 10.6 (1.95)
Statistical Analysis 1: Comparison: Treatment I: (DR-102) vs Treatment II; Test type: Superiority or Other; p = 0.8507, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares mean difference: Treatment I - Treatment II; Least Squares Mean Difference = 0.5, 95% CI 2-sided [-4.87 to 5.91]

9. Secondary Outcome: Least Squares Mean Change From Baseline Over the 6-Month Treatment Period in Activated Partial Thromboplastin Time (APTT)-Based Activated Protein-C (APC) Resistance
Description: This hemostatic parameter is calculated by dividing the clotting time with APC by the clotting time without APC. Normal range for this measure was defined as a ratio of 2.00 to 3.36. Participants were in a fasting state and had refrained from moderate to vigorous exercise prior to phlebotomy on the day of this lab draw. Change from baseline was analyzed using a repeated measures analysis of covariance with covariate adjustment for baseline, treatment, month, and the treatment by month interaction.
Time Frame: Baseline through Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Treatment I: (DR-102) | Treatment II
Number analyzed (Participants) | 124 | 120
ratio | -0.3 (0.02) | -0.4 (0.02)
Statistical Analysis 1: Comparison: Treatment I: (DR-102) vs Treatment II; Test type: Superiority or Other; p = 0.0459, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares mean difference: Treatment I - Treatment II; Least Squares Mean Difference = 0.1, 95% CI 2-sided [0.00 to 0.14]

10. Secondary Outcome: Least Squares Mean Change From Baseline Over the 6-Month Treatment Period in Endogenous Thrombin Potential (EPT)-Based Activated Protein-C (APC) Resistance
Description: This hemostatic parameter is calculated by dividing the clotting time with APC by the clotting time without APC. Normal range for this measure was defined as a ratio of 0.32 to 1.79. Participants were in a fasting state and had refrained from moderate to vigorous exercise prior to phlebotomy on the day of this lab draw. Change from baseline was analyzed using a repeated measures analysis of covariance with covariate adjustment for baseline, treatment, month, and the treatment by month interaction.
Time Frame: Baseline through Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Treatment I: (DR-102) | Treatment II
Number analyzed (Participants) | 124 | 121
ratio | 0.8 (0.04) | 0.7 (0.04)
Statistical Analysis 1: Comparison: Treatment I: (DR-102) vs Treatment II; Test type: Superiority or Other; p = 0.0318, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares mean difference: Treatment I - Treatment II; Least Squares Mean Difference = 0.1, 95% CI 2-sided [0.01 to 0.26]

11. Secondary Outcome: Least Squares Mean Change From Baseline Over the 6-Month Treatment Period in Corticosteroid-Binding Globulin
Description: Normal range for this adrenal parameter was 1906.448 to 4520.504 mg/L. Change from baseline was analyzed using a repeated measures analysis of covariance with covariate adjustment for baseline, treatment, month, and the treatment by month interaction.
Time Frame: Baseline through Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Treatment I: (DR-102) | Treatment II
Number analyzed (Participants) | 122 | 117
mg/L | 4083.3 (159.45) | 3721.8 (162.95)
Statistical Analysis 1: Comparison: Treatment I: (DR-102) vs Treatment II; Test type: Superiority or Other; p = 0.1148, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares mean difference: Treatment I - Treatment II; Least Squares Mean Difference = 361.6, 95% CI 2-sided [-88.45 to 811.61]

12. Secondary Outcome: Least Squares Mean Change From Baseline Over the 6-Month Treatment Period in Serum Random Total Cortisol
Description: Normal range for this adrenal parameter was 85.6 to 618.2 nmol/L. Change from baseline was analyzed using a repeated measures analysis of covariance with covariate adjustment for baseline, treatment, month, and the treatment by month interaction.
Time Frame: Baseline through Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Treatment I: (DR-102) | Treatment II
Number analyzed (Participants) | 125 | 120
nmol/L | 239.0 (15.67) | 230.8 (16.03)
Statistical Analysis 1: Comparison: Treatment I: (DR-102) vs Treatment II; Test type: Superiority or Other; p = 0.7136, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares mean difference: Treatment I - Treatment II; Least Squares Mean Difference = 8.2, 95% CI 2-sided [-35.92 to 52.39]

13. Secondary Outcome: Least Squares Mean Change From Baseline Over the 6-Month Treatment Period in Thyroid-Stimulating Hormone (TSH)
Description: Normal range for this parameter was 0.35 to 5.5 mIU/L. Change from baseline was analyzed using a repeated measures analysis of covariance with covariate adjustment for baseline, treatment, month, and the treatment by month interaction.
Time Frame: Baseline through Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mIU/L
Arm/Group | Treatment I: (DR-102) | Treatment II
Number analyzed (Participants) | 125 | 120
mIU/L | 0.2 (0.07) | 0.3 (0.07)
Statistical Analysis 1: Comparison: Treatment I: (DR-102) vs Treatment II; Test type: Superiority or Other; p = 0.3903, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares mean difference: Treatment I - Treatment II; Least Squares Mean Difference = -0.1, 95% CI 2-sided [-0.29 to 0.11]

14. Secondary Outcome: Least Squares Mean Change From Baseline Over the 6-Month Treatment Period in Sex Hormone Binding Globulin
Description: Normal range for this parameter was 28 to 146 nmol/L. Change from baseline was analyzed using a repeated measures analysis of covariance with covariate adjustment for baseline, treatment, month, and the treatment by month interaction.
Time Frame: Baseline through Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Treatment I: (DR-102) | Treatment II
Number analyzed (Participants) | 125 | 120
nmol/L | 163.4 (7.29) | 149.1 (7.46)
Statistical Analysis 1: Comparison: Treatment I: (DR-102) vs Treatment II; Test type: Superiority or Other; p = 0.1731, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares mean difference: Treatment I - Treatment II; Least Squares Mean Difference = 14.3, 95% CI 2-sided [-6.29 to 34.80]

ADVERSE EVENTS:
Time Frame: Adverse events/serious adverse events were collected from the time of signed informed consent until the the Final Telephone Contact (14 days after completing investigational product) or the Early Termination Visit. Treatment period was 6 28-day cycles.
Arm/Group | Treatment I: (DR-102) | Treatment II
Serious Adverse Events (participants affected / at risk) | 0/145 | 1/142
Other Adverse Events (participants affected / at risk) | 84/145 | 66/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment I: (DR-102) (N=145) | Treatment II (N=142)
Appendicitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment I: (DR-102) (N=145) | Treatment II (N=142)
Nausea (Gastrointestinal disorders) | 4 | 2
Nasopharyngitis (Infections and infestations) | 3 | 3
Gastroenteritis (Infections and infestations) | 1 | 4
Influenza (Infections and infestations) | 1 | 4
Urinary tract infection (Infections and infestations) | 1 | 3
Alpha globulin increased (Investigations) | 11 | 8
Prothrombin level increased (Investigations) | 8 | 7
Antithrombin III decreased (Investigations) | 1 | 3
Headache (Nervous system disorders) | 9 | 16
Dizziness (Nervous system disorders) | 4 | 0
Libido decreased (Psychiatric disorders) | 3 | 1
Metrorrhagia (Reproductive system and breast disorders) | 50 | 28
Breast pain (Reproductive system and breast disorders) | 5 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 4 | 7
Menorrhagia (Reproductive system and breast disorders) | 4 | 1
Amenorrhoea (Reproductive system and breast disorders) | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Acne (Skin and subcutaneous tissue disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator/Institution must submit proposed publication to Sponsor for review within a prespecified number of days before submission for publication. If Sponsor's review shows that potentially patentable subject matter would be disclosed, publication/public disclosure shall be delayed to enable Sponsor, or Sponsor's designees, to file necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.